CLINICAL TRIAL: NCT05079711
Title: Comparative Performance of the SavvyCheck Vaginal Yeast Test Versus Culture
Brief Title: Comparative Performance of a Vaginal Yeast Test
Status: Recruiting | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Savvyon Diagnostics Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: USUHS.2020-058
Record Dates: First submitted 2021-06-30; First posted 2021-10-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Vaginal candidiasis, Vaginal yeast culture
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Five vaginal swabs; one collected by the subject and four collected by a healthcare provider (healthcare provider only will use a swab randomization scheme). The five swabs will be analyzed by:
  * Vaginal wet mount microscopy (1 swab)
  * Reference Method (vaginal Candida yeast culture) (1 swab)
  * Subject and trained user-performed SavvyCheck Vaginal Yeast Test (2 swabs; 1 each)
  * PCR and sequencing of fungi (1 swab; analysis to be conducted in discordant cases only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic for vaginal yeast: Women presenting to the clinic with symptoms of vulvovaginal candidiasis.
  Interventions: Device: SavvyCheck Vaginal Yeast Test (rapid, point-of-care diagnostic test)
- Asymptomatic for vaginal yeast: Women presenting to the clinic with no symptoms of vulvovaginal candidiasis.
  Interventions: Device: SavvyCheck Vaginal Yeast Test (rapid, point-of-care diagnostic test)

INTERVENTIONS:
Device: SavvyCheck Vaginal Yeast Test (rapid, point-of-care diagnostic test) — The SavvyCheck Vaginal Yeast Test is a lateral flow immunochromatographic qualitative test for detection of Candida antigen in vaginal secretions, sampled by a swab as an aid for identification of vulvovaginal candidiasis (VVC), as a primary cause of vaginal yeast infections. The SavvyCheck Vaginal Yeast Test is designed for use by women experiencing vaginal symptoms, including: increased vaginal discharge, vaginal itching, vaginal soreness and irritation, rash on the labia, and genital burning that may worsen during urination. The SavvyCheck Vaginal Yeast Test is indicated for OTC use.

SUMMARY:
The purpose of this study is to establish lay user performance criteria for the SavvyCheck Vaginal Yeast Test in comparison to standard vaginal yeast culture and identification method for Candida (the Reference Method). Polymerase chain reaction (PCR) and sequencing of fungi will be used as an aid to explain the nature of the discrepancy in the case of discordant results between the lay user-performed SavvyCheck Vaginal Yeast Test and standard vaginal yeast culture and identification method for Candida.

DETAILED DESCRIPTION:
The purpose of this study is to establish lay user performance criteria for the SavvyCheck Vaginal Yeast Test in comparison to standard vaginal yeast culture and identification method for Candida (the Reference Method). Polymerase chain reaction (PCR) and sequencing of fungi will be used as an aid to explain the nature of the discrepancy in the case of discordant results between the lay user-performed SavvyCheck Vaginal Yeast Test and standard vaginal yeast culture and identification method for Candida.

Primary Objective:

The primary objective is to establish lay user performance criteria (sensitivity and specificity) of the SavvyCheck Vaginal Yeast Test in comparison to the Reference Method (vaginal Candida yeast culture)

Secondary Objectives:

1. To determine the positive predictive value and negative predictive value of the lay user-performed SavvyCheck Vaginal Yeast Test in comparison to the Reference Method (vaginal Candida yeast culture)
2. To determine the concordance between the results determined by lay user-performed SavvyCheck Vaginal Yeast Test -vs. trained user-performed SavvyCheck Vaginal Yeast Test

Exploratory Objectives:

1. To determine the concordance between the results determined by lay user-performed SavvyCheck Vaginal Yeast Test -vs. vaginal wet mount microscopy results
2. To determine the concordance between results determined by lay user-performed SavvyCheck Vaginal Yeast Test -vs. PCR and sequencing
3. To determine the concordance between results determined by the Reference Method (vaginal Candida yeast culture) -vs. PCR and sequencing

Primary Endpoints:

Calculation of sensitivity and specificity of the lay user-performed SavvyCheck Vaginal Yeast Test as compared to the Reference Method (vaginal Candida yeast culture)

Secondary Endpoints:

1. Calculation of positive and negative predictive value of lay user-performed SavvyCheck Vaginal Yeast Test results as compared to the Reference Method (vaginal Candida yeast culture)
2. Calculation of concordance between the results determined by lay user-performed SavvyCheck Vaginal Yeast Test results -vs. trained user-performed SavvyCheck Vaginal Yeast Test results

Exploratory Endpoints:

1. Calculation of concordance between the results determined by lay user-performed SavvyCheck Vaginal Yeast Test -vs. vaginal wet mount microscopy
2. Calculation of concordance between results determined by lay user-performed SavvyCheck Vaginal Yeast Test -vs. PCR and sequencing
3. Calculation of concordance between results determined by the Reference Method (vaginal Candida yeast culture) -vs. PCR and sequencing

Women, aged 18 years and older, symptomatic and asymptomatic for vaginitis will be enrolled in the study. We estimate that it will require a total enrollment of up to 600 symptomatic women at all clinical sites combined, to achieve the target of at least n=216 Reference Method (vaginal Candida yeast culture) positives. In addition, a combined total of 320 asymptomatic women will be enrolled in the study from the four clinical sites combined, to achieve the target of at least n=170 Reference Method (vaginal Candida yeast culture) negatives.

Three, large, regional, DoD military treatment facilities (MTFs)

1. Womack Army Medical Center (WAMC) at Fort Liberty; Fayetteville, NC
2. Landstuhl Regional Medical Center (LRMC); Landstuhl, Germany
3. Brooke Army Medical Center (BAMC); Fort Sam Houston, TX

The SavvyCheck Vaginal Yeast Test is a lateral flow immunochromatographic qualitative test for the detection of Candida antigen in vaginal secretions sampled by a swab, as an aid for identification of vulvovaginal candidiasis as a primary cause of vaginal yeast infections. The SavvyCheck Vaginal Yeast Test is designed for use by women experiencing vaginal symptoms, including: increased vaginal discharge, vaginal itching, vaginal soreness and irritation, rash on the labia, and genital burning that may worsen during urination. The SavvyCheck Vaginal Yeast Test is indicated for over-the-counter use.

ELIGIBILITY:
Inclusion Criteria:

Symptomatic Women Symptomatic women include those women who present with a complaint consistent with symptoms of vaginitis (e.g., increased vaginal discharge, vaginal itching, vaginal soreness and irritation, rash on the labia, and genital burning that may worsen during urination). Enrollment will continue at each clinical site until our target number of 216 Reference Method (vaginal Candida yeast culture) positives have been collected. We estimate up to 600 symptomatic women will be enrolled to meet our target.

Inclusion Criteria for Symptomatic Women

1. DoD Military Health System beneficiary
2. Have a healthcare appointment at a recruitment clinic
3. 18 years of age or older
4. Must speak and understand English
5. Able to provide informed consent
6. Women experiencing vaginal symptoms, including: increased discharge, itching, soreness and irritation, rash on the labia, and genital burning that may worsen during urination
7. Must determine the test is applicable to her based on her symptoms after she has read the outside device labeling (box label)

Asymptomatic Women Asymptomatic women include those women who do not present with a complaint consistent with vaginitis. Enrollment will continue at each clinical site until our target number of 170 Reference Method (vaginal Candida yeast culture) negatives have been collected. We estimate up to 320 asymptomatic women will be enrolled to meet our target.

Inclusion Criteria for Asymptomatic Women:

1. DoD Military Health System beneficiary
2. Have a healthcare appointment at a recruitment clinic
3. 18 years of age or older
4. Must speak and understand English
5. Able to provide informed consent
6. Healthy women appearing for routine care without symptoms of vaginal yeast infection

Exclusion Criteria:

If any of the following criteria are met, a potential subject will be excluded from the study:

1. Currently menstruating
2. History of any clinical therapies and/or interventions related to gender confirmation (transgender person)
3. Use of any vaginal medication, taken by mouth or vaginally, within the last 7 days
4. Use of any vaginal product within 24 hours, including contraception (cream, gel, or foam), or douching solutions

NOTE: Women who currently have an intrauterine device (IUD) placed are eligible to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women experiencing vulvovaginal symptoms of candidiasis vaginitis.
Study Population: Women, aged 18 years and older, symptomatic and asymptomatic for vaginitis will be enrolled in the study. We estimate that it will require a total enrollment of up to 600 symptomatic women at all clinical sites combined, to achieve the target of at least n=216 Reference Method (vaginal Candida yeast culture) positives. In addition, a combined total of 320 asymptomatic women will be enrolled in the study from the four clinical sites combined, to achieve the target of at least n=170 Reference Method (vaginal Candida yeast culture) negatives.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Assess sensitivity and specificity between lay user-performed SavvyCheck Vaginal Yeast Test result compared to the Reference Method (vaginal Candida yeast culture) | 12 months
  Calculation of sensitivity and specificity of the lay user-performed SavvyCheck Vaginal Yeast Test as compared to the Reference Method (vaginal Candida yeast culture)

SECONDARY OUTCOMES:
Assess positive and negative predictive values of the lay-user SavvyCheck Vaginal Yeast Test result as compared to the Reference Method (vaginal Candida yeast culture) | 12 months
  Calculation of the positive and negative predictive values of lay user-performed SavvyCheck Vaginal Yeast Test results as compared to the Reference Method (vaginal Candida yeast culture).
Assess concordance between the lay user-performed SavvyCheck Vaginal Yeast test result and the trained user-performed result. | 12 months
  Calculation of concordance between the lay use-performed and the trained user-performed SavvyCheck Vaginal Yeast test results.

OTHER OUTCOMES:
Assess concordance between the lay user-performed SavvyCheck Vaginal Yeast test result -vs vaginal wet mount microscopy | 12 months
  Calculation of concordance between the results between the lay user-performed SavvyCheck Vaginal Yeast Test -vs. vaginal wet mount microscopy
Assess concordance between the lay user-performed SavvyCheck Vaginal Yeast test result -vs. PCR and sequencing | 12 months
  Calculation of concordance between the results between the lay user-performed SavvyCheck Vaginal Yeast Test -vs. PCR and sequencing
Assess concordance between the Reference Method results (vaginal yeast culture) -vs PCR and sequencing | 12 months
  Calculation of concordance between the Reference Method (vaginal yeast culture) results -vs PCR and sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Kostas-Polston, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (3):
- United States (2):
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
- Landstuhl Regional Medical Center, Landstuhl, Germany

IPD SHARING:
Plan to Share IPD: No